CLINICAL TRIAL: NCT02933138
Title: Systematic Study of Post Herapin Lipoprotein Lipase Activity and Lipoprotein Remodelling in Multifactorial Chylomicronemia
Brief Title: Plasma Triglyceride Lipolysis in Multifactorial Chylomicronemia
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0636
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Hyperlipoproteinemia
Keywords: Lipoprotein Lipase; Hypertriglyceridemia; Triglycerides; Lipolysis; Multifactorial Chylomicronemia
MeSH Terms: conditions — Hyperlipoproteinemias; Hypertriglyceridemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — post-heparin EDTA plasma ADN

GROUPS / COHORTS (1):
- Multifactorial Chylomicronemia: no intervention, phenotypic and genotypic study

SUMMARY:
Purpose: The mechanism of most of the multifactorial chylomicronemia (MCM) remains elusive. In order to decipher the mechanisms involved in the occurrence of this disease, plasma TG lipolysis characteristics will be monitored for 60 minutes after heparin injection instead of the 10 minutes gold standard, in a large group of genotyped MCM patients.

DETAILED DESCRIPTION:
Purpose: The mechanism of most of the multifactorial chylomicronemia (MCM) remains elusive. In order to decipher the mechanisms involved in the occurrence of this disease, plasma TG lipolysis characteristics will be monitored for 60 minutes after heparin injection instead of the 10 minutes gold standard, in a large group of genotyped MCM patients.

Method: LPL, APOC2, APOA5, GPIHB1and APOE genotypes will be determined for each patient. Basal lipid profiles including Apo B, CII, CIII, and lipoprotein lipase (LPL) concentration will be measured in 62 MCM patients, in addition to LPL activity (PHLA) T0, T10 T30 T60 minutes, Assessment of TG chylomicron decrease Study of lipoprotein remodelling by agarose gel electrophoresis.

Hypothesis To confirm the preliminary finding of high LPL activity in multifactorial chylomicronemia To explore the interest of a longer assessment of LPL activity following heparin injection. To establish if specific phenotypes could be identified among MCM patient supporting the hypothesis of different mechanisms involved (ie overproduction or defect in hepatic clearance)

ELIGIBILITY:
Inclusion Criteria:

* patient with a documented history of MCM (Plasma TG concentration (TG) > 15 mmol/l or familial history of hypertriglyceridemia with TG >10 mmol/l)
* no contraindication for a single heparin injection for ex vivo LPL activity assessment

Exclusion Criteria:

* patients carriers of homozygous or compound heterozygous mutations on LPL, GPIHBP1, APOA5, APOC2 or APOE genes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with a documented history of MCM (Plasma TG concentration (TG) > 15 mmol/l or familial history of hypertriglyceridemia with TG >10 mmol/l) who had no contraindication for a single heparin injection for ex vivo LPL activity assessment
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2010-07; Primary Completion 2012-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Lipoprotein Lipase concentration | 60 minutes after heparin injection

SECONDARY OUTCOMES:
Basal lipid profiles | maximum 60 min before heparin injection
Lipoprotein electrophoresis | maximum 60 minutes after heparin injection
Total triglycerides decrease | maximum 60 minutes after heparin injection